CLINICAL TRIAL: NCT07226739
Title: Comprehensive Toileting Programming: Enuresis Treatment to a Randomized Clinical Trial of a Caregiver-Mediated Multidisciplinary Intervention for Encopresis
Brief Title: Comprehensive Toileting Program
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mindy Scheithauer, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00010223; 1R01HD115933-01A1 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Encopresis; ASD
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded independent evaluator will conduct the Clinical Global Impression scale.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caregiver-mediated version of multidisciplinary intervention for encopresis (CM-MIE) Arm (Experimental): * A Board-Certified Behavior Analyst (BCBA) will meet virtually with caregivers for daily appointments for two weeks (goal of 10 appointments; maximum of 2-hours per appointment).
  * First appointment, the BCBA will provide support on using telehealth and psychoeducation about encopresis, reinforcement, and suppository use.
  * Subsequent appointments involve a scheduled sit on the toilet to encourage an independent bowel movement. If a bowel movement occurs, the caregiver is coached to provide the child with a highly preferred item, praise, and allow them to leave the bathroom. If a bowel movement does not occur, the therapist coaches the parent through administration of a glycerin suppository intended to quickly elicit a bowel movement, followed by another scheduled sit on the toilet.
  * After consistent success with continent BMs following suppository administration, the suppository dose will be reduced to gradually fade out its use.
  Interventions: Drug: Glycerin Suppository; Behavioral: Behavioral strategies
- Parent Education (PE) Arm (Active Comparator): * PE includes an initial appointment with a BCBA who will provide recommendations on promoting bowel movement continence.
  * First appointment will involve a didactic review of the basics of reinforcement, collecting data to identify when BMs are most likely, and scheduled sits around this time. Caregivers will be instructed to collect data on BMs after this appointment.
  * The BCBA will then hold daily follow-up appointments (10 appointments total over 2 weeks). At these appointments, the BCBA will review this data and make additional recommendations (e.g., changing the timing of scheduled sits based on when BMs are most likely to occur, altering the reinforcer used for continent voids) to promote success.
  Interventions: Behavioral: Behavioral strategies

INTERVENTIONS:
Drug: Glycerin Suppository — Liquid glycerin suppositories, pediatric (age 2-5 years: 4 ml/applicator) or adult (6-12 years: 7.5ml/applicator) dose used as indicated based on age will be used in the study. Up to two doses will be delivered a day.
  The purpose of the glycerin suppository is to rapidly evoke a bowel movement, which allows for a predictable bowel movement to occur while the child is seated on the toilet (a continent bowel movement).
  Other Names: MAJOR® Glycerin
  Arms: Caregiver-mediated version of multidisciplinary intervention for encopresis (CM-MIE) Arm
Behavioral: Behavioral strategies — The BCBA will provide recommendations on promoting bowel movement continence. The caregiver will be asked to collect data between visits that will be reviewed by the therapist.

SUMMARY:
The current study aims to monitor fecal continence after autistic youth complete enuresis treatment and for individuals who continue to experience encopresis after acquiring urine continence, evaluate a caregiver-mediated version of a Multidisciplinary Intervention for Encopresis (CM-MIE) delivered via telehealth to determine efficacy in a randomized clinical trial.

DETAILED DESCRIPTION:
Participants will complete toilet training for enuresis (if needed) and then monitored to determine if encopresis persists. For individuals with resolved enuresis but persisting encopresis, they will be randomized to receive either a treatment for encopresis (delivered via telehealth) or a parent education program. The encopresis intervention involves behavioral components and administration of an over-the-counter suppository as needed. All participants will also meet with a pediatric gastroenterologist to ensure safety of study procedures and to resolve constipation as needed. Outcomes will include caregiver-completed questionnaires, data on bowel movements collected by the caregiver, and an interview between the participant's caregiver and a blinded investigator focused on encopresis, other presenting concerns, and any potential adverse events.

Informed consent will be collected via signature from one legal guardian. The investigators will collect assent from participants when appropriate given age and developmental level.

ELIGIBILITY:
Inclusion Criteria

* Age 5 to 12
* Diagnosis of an intellectual or developmental delay (excluding individuals with ADHD alone)
* Encopresis (more than 1 incontinent BM a week)
* Required for pre-randomization phase only: Enuresis (> 1 incontinent urination per day when on a consistent toileting sit schedule)
* At least one caregiver who speaks and understands English

Exclusion Criteria:

* Unresolved medical condition that would impede toilet training (e.g., interference with sphincter control, short gut syndrome, urinary tract or gastrointestinal infection, unexplained diarrhea, recent intestinal surgery, inflammatory bowel disease)
* Failed intensive toileting treatment in the past 2 yrs with protocols akin to study
* Current serious behavioral or psychiatric disorder that requires another treatment
* Current or planned other intervention (behavioral or medical) for incontinence

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Improvement (CGI-I) scale score | 5 weeks post-baseline (Endpoint)
  The CGI-I is a clinician-rated 7-point scale measuring overall change from baseline. Scores range from 1 (Very Much Improved) to 4 (Unchanged) to 7 (Very Much Worse), rated by the treatment-blind independent evaluator (IE) with all available information. CGI-I ratings of Much Improved (score of 2) or Very Much Improved (score of 1) will define positive response; all other ratings are defined as nonresponders. Number of positive responses for the Clinical Global Impression scale will be compared between the CM-MIE and the PE group.

SECONDARY OUTCOMES:
Caregiver Strain Questionnaire-short form (CGSQ-SF) score | 5 weeks post-baseline (Endpoint)
  Caregiver Strain Questionnaire-short form (CGSQ-SF) change score at endpoint will be compared between the CM-MIE and the PE group.
  The Caregiver Strain Questionnaire-short form is a 7-item measure of self-reported strain experienced by caregivers and families, with responses on a 5-point Likert scale. Total possible score range is 7-35, with higher scores indicating higher strain (worse outcome).
Fecal continence based on caregiver-collected data | 5 weeks post-baseline (Endpoint)
  Treatment response measured as fecal continence based on caregiver-collected data in a bowel-activity diary that documents all continent and incontinent bowel movements. Number of positive responses will be compared in CM-MIE vs. PE groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Scheithauer, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The below information will all be shared through NIMH Data Archive (NDA):
  1. Diagnostic information
  2. Scores from developmental measures (e.g., ADOS or CARS)
  3. Vineland Adaptive Behavior Scale
  4. Differential Ability Scale or Mullen Scales of Early Learning
  5. Aberrant Behavior Checklist
  6. Caregiver Strain Questionnaire
  7. Open Source - Challenging Behavior Checklist
  8. Clinical Global Impression scale (Improvement Scale)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be submitted via the time standards set forth by NDA.
Access Criteria: Access to data for research purposes will be provided through an NDA Data Access Committee (DAC). Investigators and institutions seeking data from NDA will be expected to meet data security measures and will be asked to submit a Data Use Certification, which is cosigned by the investigator and the designated Institutional Official(s) at the NIH-recognized sponsoring institution with a current Federal Wide Assurance (FWA).